CLINICAL TRIAL: NCT05088941
Title: Impact of SARS-CoV-2 Pandemic on Allogeneic Stem Cell Transplantation Organization : a French Experience
Brief Title: Impact of COVID-19 Pandemic on Allogeneic Stem Cell Transplantation Organization : a French Experience
Acronym: covidallo
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, DECOT Véronique, professor, Central Hospital, Nancy, France
Other Study IDs: 2021PI153
Record Dates: First submitted 2021-10-15; First posted 2021-10-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Allogeneic Stem Cell Transplantation; SARS-CoV2 Infection; COVID-19
Keywords: allogeneic stem cell transplant; SARS-CoV2; freezing process
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the SARS-CoV2 pandemic has led to a major reorganization of the French Hematology and stem cell transplant departments since march 2020. Since the allogeneic stem cell transplant cannot be delayed especially when patients with hematological malignancies are in a fragile remission, risking relapse at any time, the necessity to maintain safe hematopoietic stem cell (HSC) donations from match unrelated or family donors appears rapidly mandatory during the pandemic period. To increase the safety of voluntary donations, a SARS-CoV2 Polymerase Chain Reaction test has been recommended to donors by regulatory agencies. However, due to the lack of homogeneity of care at European level, some countries do not require SARS-CoV-2 testing in asymptomatic donors. In this case, the test is performed on additional EDTA tube accompanying the graft on arrival or in the case of a missing tube (not collected or forgotten), on few milliliters of the HSC graft. This circuit had the consequence of forcing the clinicians to wait for the test result before starting the patient's conditioning regimen. The graft being already collected and received at the transplant center, and the conditioning regimen lasting on an average of 5 days, this resulted in its conservation during this minimum period and therefore its freezing by the associated cell therapy unit. However, this practice has so far been exceptional regarding allogeneic transplants, which are primarily freshly infused to ensure to the recipient the highest viability and functionality of stem cells. Since the entire freezing-thawing and washing process may impact cell viability and delay the patient's aplastic recovery, this study aimed to analyze the results of one year of allogeneic transplants infused after freezing in terms of graft quality after thawing and clinical consequences.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving an allogeneic stem cell transplant between march 2020 and may 2021.

Exclusion Criteria:

* patients receiving an allogeneic stem cell transplant before march 2020 and after may 2021.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (children and adults) having HSCT and treated at the CHRU of NANCY between march march 2020 to may 2021
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
% of Total Nucleated Cell (TNC) yield (final TNC count / initial TNC count) | 2020-2021
%of CD34 + cells yield (final CD34+ cell count / initial CD34+ cell count) | 2020-2021
% of CFU-GM yield (final CFU-GM count / initial CFU-GM count) | 2020-2021
% of post-thaw CD34 viability | 2020-2021
% of post-thaw TNC viability | 2020-2021

SECONDARY OUTCOMES:
GvHD incidence | 2020-2021
infections rate | 2020-2021
relapse rate | 2020-2021
death rate | 2020-2021
graft rejection | 2020-2021
aplastic recovery | 2020-2021

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU of Nancy, Vandœuvre-lès-Nancy, Meurthe-et-Moselle, France